CLINICAL TRIAL: NCT05507866
Title: Evaluation of a Comprehensive School Nutrition Enrichment Intervention (CSNEI) in Rural School Districts
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 273437
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Obesity, Childhood; Nutrition, Healthy
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Matched-pairs cluster-randomized trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSNEI (Experimental): Schools randomized to receive the CSNEI intervention arm will receive help in addressing childhood obesity by modifying meal/menu items, changing school cafeteria environments, and making changes to purchasing and procurement practices.
  Interventions: Other: CSNEI
- Control (No Intervention): Schools randomized to the control arm will follow their existing nutritional practices.

INTERVENTIONS:
Other: CSNEI — CSNEI is a policy intervention designed to address childhood obesity by modifying lunch and breakfast meal/menu items, changing the school cafeteria environments, and making changes to purchasing and procurement practices.
  Arms: CSNEI

SUMMARY:
Obesity is a significant cause of cancer and cardiovascular disease incidence and mortality, and diabetes incidence among rural communities. Arkansas has the sixth-highest proportion of rural population (~41%),and has the third-highest obesity prevalence (37.4%) in the nation. Arkansas has the third-highest prevalence of obesity for high school students (22.1%) and the fifth-highest prevalence for children ages 10-17 (20.2%). In Arkansas, children in rural areas have very high rates of both food insecurity (26%) and free and reduced lunch eligibility (72.9%). In the study's 6 participating school districts, free and reduced lunch eligibility ranges from 51.4% to 79.3%. School meals are an important opportunity to influence students' nutritional intake and long-term food preferences, which can reduce obesity. A multidisciplinary team partnered with 6 rural Arkansas school districts which to evaluate the effects of an evidence-based population-level intervention designed to improve the nutritional quality of food served in schools.

The primary research question is: "Compared with similar school districts that did not implement the CSNEI, does the CSNEI intervention yield improved obesity prevention outcomes among rural K-12 students?" The study team will conduct a matched-pairs cluster-randomized trial with pre-test and repeated post-tests in 6 rural Arkansas school districts, 3 implementing CSNEI, and 3 matched comparison school districts following their existing nutritional practices. The evaluation will include ~11,500 students in 6 school districts: ~5,750 from CSNEI school districts and ~5,750 from matched comparison school districts. The study will explore heterogeneity of treatment effects for age and economic standing to understand effects on populations with higher contextual risk for obesity. Baseline data collection will take place prior to implementation (Year 1), and follow-up data will be collected annually thereafter (Years 2-4). The specific aims are: Aim 1.A: Evaluate the effects of a CSNEI on students' relative BMI change over time. Aim 1.B: Evaluate the short-term and long-term effects of a CSNEI on the nutritional quality of food served in school meals. Aim 1.C: Evaluate the short-term and long-term effects of a CSNEI on students' consumption of food served in school meals. Aim 1.D: Evaluate the short-term and long-term effects of a CSNEI on students' skin carotenoid levels, as an indicator of fruit and vegetable intake.

ELIGIBILITY:
Inclusion Criteria:

- Student currently enrolled at one of the 6 rural public school districts

Exclusion Criteria:

- N/A

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11536 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in student body mass index (BMI) z-score | Baseline; 3 years post-intervention; 5 years post-intervention
  Student BMI data will be provided by the Arkansas School BMI Database. Changes in BMI z-score will be assessed from baseline to each follow-up time point.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Long, PhD, Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences Northwest, Springdale, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No